CLINICAL TRIAL: NCT07267429
Title: Resistance Training-induced Adaptations in Children
Acronym: B-STRONG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Bareket Falk, Professor, Brock University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B-STRONG
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: Strength training; Resistance training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Active Comparator): resistance training, 12 weeks, 2 times per week
  Interventions: Other: Resistance training
- Control (No Intervention): continue with habitual physical activity

INTERVENTIONS:
Other: Resistance training — progressive resistance training, 12 weeks, 2 times per week
  Arms: Training

SUMMARY:
Resistance exercise training (RET) in children and adolescents has become a popular activity, with a growing body of evidence supporting its use. Numerous studies indicate that it is safe and effective at increasing muscular strength, improving sport performance, and mitigating injury risk. Despite this evidence, there are still many unknowns with RET in children, including its mechanisms of action in enhancing muscle strength.

Neural and muscular mechanisms can improve muscle strength following RET. Neural factors include improved recruitment and firing of an individual's muscle cells, and muscular factors primarily include an increase in the size of the muscle (hypertrophy). In children, little is known about how these mechanisms relate to muscle strength.

Therefore, the purpose of this study is to non-invasively assess the mechanisms of RET-induced strength increases in children performing 12 weeks of RET, compared with a non-training control group. Broadly, muscular adaptations will be assessed using ultrasound measures, while neural mechanisms will be assessed using surface electromyography decomposition.

DETAILED DESCRIPTION:
Resistance exercise training (RET) in children and adolescents has become a popular activity, with a growing body of evidence supporting its use. Position and consensus statements on RET for children indicate that it is safe and effective at increasing muscular strength, improving sport performance, and mitigating injury risk. Despite this evidence, there are still many unknowns with RET in children, including its mechanisms of action in enhancing muscle strength.

Neural and muscular mechanisms can improve muscle strength following RET. Neural factors include improved recruitment and firing of an individual's motor units, and muscular factors primarily include an increase in the size of the muscle (hypertrophy). In children, little is known about how these mechanisms relate to muscle strength. There is very little evidence of morphological changes following RET in children. Therefore, conventional wisdom is that children rely only on neural factors to improve strength following RET, possibly due to their lower levels of circulating androgens. Nevertheless, some studies have suggested RET-induced muscle hypertrophy in children and adolescents, indicating that with certain training protocols, and with more-sensitive research methods, children may achieve RET-induced muscle growth.

The neural mechanisms that presumably improve the muscle strength of children following RET are also largely unknown. Previously, global surface electromyography (sEMG) has been utilized to observe changes in overall muscle activation. However, this measure is unspecific and can be influenced by neural and morphological adaptations. Recent advancements in sEMG decomposition - which separates the sEMG signal into the discrete motor units it is composed of - allow for more specific neural adaptations to be assessed non-invasively. To date, this technological advancement has only been utilized in two studies to assess neuromuscular adaptations to RET in youths, with inconsistent results.

Therefore, the purpose of this study is to non-invasively assess the mechanisms of RET-induced strength increases in children performing 12 weeks of RET, compared with a non-training control group. Broadly, morphological adaptations will be assessed using ultrasound measures, while neural mechanisms will be assessed using sEMG decomposition. In addition to these primary outcomes, the effects of RET in children on cardiovascular regulation.

Procedures Participants will be required to make three pre-intervention, two mid-intervention, and two post-intervention visits to the Applied Physiology/Sympathetic Neurocirculatory Regulation Laboratories at Brock University for the completion of all testing procedures. The mid-intervention visits will be during the fourth and eighth weeks (1 session each), and the post intervention visits will be within one week following the completion of the intervention (2 sessions).

The first pre-intervention visit will serve as the familiarization session. Questionnaires will be completed to screen for medical concerns, assess pubertal stage, athletic training practices, menarcheal status (females only), self perception, habitual eating habits, and habitual physical activity. These questionnaires will be repeated following the intervention period. Following the completion of questionnaires, participants will be familiarized with the muscular strength/contraction tests that will be performed in the remaining testing sessions.

Four of the remaining testing sessions (1 pre-intervention, 2 mid-intervention, and 1 post-intervention) will include body measures and muscular strength/contraction tests that will serve as the primary experimental outcomes. Finally, one of the pre- and post-intervention sessions will include the assessment of blood flow and pressure regulation, to see how these are affected by RET.

The RET protocol will include twice weekly RET sessions for 12 weeks, using exercise machines. Each session will consist of ~5-10 minutes of warm-up, ~40-50 minutes of resistance training exercises, and ~5-10 minutes of cool down. The program will primarily focus on exercise machines for the lower body; however, some free weight and upper body exercises will be incorporated to maintain the interest of the participants and to ensure a whole-body workout. Exercises will be completed at varying intensities and volumes, but generally between 60-85% 1RM for ~6-15 repetitions. When the desired number of repetitions can be performed by a participant safely and with appropriate technique, the intensity (e.g., weight) of the exercise will be progressed. Some examples of exercise that will be of focus in the training protocol will include the leg press, leg extension, and leg curl. Prior to the administering the intervention, participants will be properly shown how to safely conduct each exercise in a controlled and safe manner.

Participants in the proposed study will be male and female children (~7-12 years).

ELIGIBILITY:
Inclusion Criteria:

* healthy
* able to exercise

Exclusion Criteria:

* have consumed any medications in the past year which may affect muscle function,
* have any prior injuries or medical diagnoses associated with altered muscular function,
* have had an injury in the past 6 months that would limit the movements required for the training and assessment protocols,
* have performed resistance training in the past 6 months or currently participate in competitive sports (i.e., outside of school) more than 2x/week.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
muscle strength | From enrollment to the end of training at 12 weeks
  1 repetition maximal - knee extension
Peak torque | From enrollment to end of training at 12 weeks
  Peaktorque will be measured during isokinetic and isometric maximal contractions of the knee extensors

SECONDARY OUTCOMES:
Motor unit activation | from enrollment to end of training at 12 weeks
  Surface electromyography signal during a ramped contraction will be used to assess changes in motor unit firing rates
muscle cross sectional area | from enrollment to end of training at 12 weeks
  B-mode ultrasound will be used to capture panoramic images of multiple muscles of the thigh. These images will be used to assess changes in muscle cross sectional area.
Blood pressure regulation | from enrollment to end of training at 12 weeks
  Blood pressure will be assessed before and after maximal voluntary apnea, as well as before and after isometric handgrip exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Bareket Falk, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, Saint Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Participation is confidential